CLINICAL TRIAL: NCT03234218
Title: Vitamin D Levels in Liver Transplantation Recipients Prospective Observational Study
Acronym: D-LIVER-X
Status: Completed | Type: Observational
Sponsor: The Mediterranean Institute for Transplantation and Advanced Specialized Therapies (Other)
Responsible Party: Sponsor
Other Study IDs: IRRB/12/16
Record Dates: First submitted 2017-07-14; First posted 2017-07-31 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2017-09

CONDITIONS: Liver Transplant Disorder; Vitamin D Deficiency
Keywords: vitamin D, liver transplantation
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Interest in vitamin D has seen an unprecedented revival sparked by the finding that vitamin D has pleiotropic effects with an intriguing link to the critically ill patients. The recent VITdAL-ICU RCT found a significant difference in mortality in patients with severe deficiency when high doses of vitamin D supplementation were administered.

Vitamin D deficiency is extremely common in patients with chronic liver disease and/or cirrhosis. It seems to be a marker of severity of the disease, but also a possible contributing factor in determining poor outcomes.

Design of the study: Observational prospective study. Primary variable end point: Vitamin D at baseline, and POD (post-operative day) 1, 3, 7, 28.

Secondary variable end points: ICU length of stay; SAPS 2 and SOFA score at POD 1, 7; Days of mechanical ventilation; Hospital length of stay; Mortality at POD 28; Diagnosed invasive infections; Graft rejection in the first 28 days; Bilirubin and INR at POD 7 and 28.

SAFETY. The patient will not undergo to additional procedure during the study and will be asked for consent to treatment of personal data.

SAMPLE SIZE. Because of the lack of knowledge in this specific cohort no formal sample was calculated beforehand. The sample size will be defined by one-year clinical activity: about 60 consecutive patients.

STATISTICAL ANALYSIS. All statistical analysis and results will be assessed and reported as exploratory analysis. In order to describe the trend over time of the vitamin D levels, descriptive statistics such as mean, median, interquartile range and standard deviation will be evaluated. In addition, 95% confidence intervals for mean and standard deviation will be reported. Comparisons between two temporal observations will be assessed with paired t-test. Any univariate association between factors or covariates, will be explored. Statistical analyses will be done with SAS 9.4,

DETAILED DESCRIPTION:
BACKGROUND Interest in vitamin D has seen an unprecedented revival sparked by the finding that vitamin D has pleiotropic effects. The nuclear vitamin D receptor (VDR) is widely present in different cell types and organs and regulates more than 200 genes.

The link between vitamin D and critical illness is new, but intriguing, because vitamin D deficiency

* has a very high prevalence in the ICU
* is strongly associated with excess morbidity and mortality
* is associated with increased susceptibility to sepsis thought its immunomodulating effects
* has a relation with acute kidney injury, acute respiratory failure, duration of mechanical ventilation and ARDS Critically ill patients are at high risk of mortality and standard care uses little or no vitamin D.

It may well be the case that vitamin D deficiency is indeed an "invisible accomplice to morbidity and mortality," as proposed by Paul Lee.

VITAMIN D IN PATIENTS WITH CHRONIC LIVER DISEASE AND/OR CIRRHOSIS Vitamin D deficiency is extremely common in patients with chronic liver disease and/or cirrhosis. It seems to be a marker of severity of the disease, but also a possible contributing factor in determining poor outcomes.

Mechanisms Low synthesis. Severe liver disease decreases vitamin D hydroxylation and albumin and DBP production. But lack of liver function is just one piece of the puzzle. Possible concomitant causes may include inadequate sun exposure, insufficient food intake, steroids, jaundice-related deterioration of vitamin synthesis on the skin, and decreased vitamin D absorption caused by intestinal edema secondary to portal hypertension or cholestasis-induced bile salt disruption.

Signaling disruption. Vitamin D plays a role in reducing risk of chronic diseases. This most likely results from local production of 1a25(OH)2D, with its autocrine and paracrine actions in cellular proliferation and differentiation. These effects may also be relevant in liver diseases.

Pro-inflammatory signals in monocytes and macrophages may regulate the local metabolism of vitamin D, and the local production of α25(OH)2D. Almost 90% of tissue macrophages are in the liver, suggesting that local production of vitamin D in liver inflammation is impaired.

Innate immunity. Vitamin D increases secretion of antibacterial proteins such as cathelicidin and beta-defensin, promotes chemotaxis and macrophage phagocytosis, and regulate the expression of several TLRs.

Adaptive immunity. Vitamin D seems to control excessive immune response by decreasing the expression of class II HLA complex, and by modulating T cells, inducing differentiation and expansion of regulatory T cells, which secrete IL-10 and TGF-β. This could explain an association between vitamin D deficiency and autoimmune liver damage. Moreover in vitro and in vivo studies of mouse models with liver fibrosis reported an anti-fibrotic effect for vitamin D.

Hepatitis C. Data have shown that vitamin D supplementation during interferon and ribavirin increased the level of sustained viral response. Furthermore, vitamin D seems to indirectly inhibit HCV replication in human hepatocytes by stimulating IFB beta production.

NAFLD. Non-alcoholic fatty liver disease is a clinical entity ranging from steatosis to non-alcoholic steatohepatitis and cirrhosis. Vitamin D deficiency has a possible role in it.

The impact of liver transplantation on vitamin D status: lack of knowledge Individual outcome after liver transplantation varies widely due to multi-factorial variables. Vitamin D has not been extensively evaluated in patients undergoing liver transplantation. In one cohort of patients, vitamin D deficiency was associated with acute cellular rejection. It is still unclear how it acts in the more critical days after transplantation, and what predictive role it may play.

The relevant role of calcium metabolism and vitamin D after solid organ transplantation has been highlighted by several meta-analyses in recent years, suggesting a possible impact on prognosis.

To stress the relevance of the topic even in such a complex surgical procedure, low vitamin D is associated with a worse outcome after various types of surgery.

Myriad considerations suggest its evaluation in liver transplantation recipients:

* Vitamin D deficiency is a global health problem.
* Patients affected with liver disease have much lower levels of vitamin D
* Causes of low levels of vitamin D may be low production, low sun exposure, reduced mobility, and other factors reducing the availability of vitamin D in the system.
* Vitamin D has pleiotropic effects, and seems to act mainly on the immunomodulating system. Infection is the main threat in the first 6 months after transplantation.
* The number of patients receiving marginal donor organs is increasing. In many of them the recovery of liver function proceeds slowly.
* Some liver recipients become severely ill during the ICU stay. In these patients there is a suspicion of severe vitamin D insufficiency.
* Incidence of acute kidney injury is very high in complicated liver transplantation.
* The VITdAL-ICU RCT found a reduced mortality in severe deficiency after high doses of vitamin D.
* Vitamin D may reveal itself as a marker of improving metabolic function, acting as a prognostic marker that may even contribute to outcome, and is easily modifiable.

Aims of the study Principal

- Describe the level and the trend of vitamin D levels in liver transplantation recipients during the first 28 days after transplantation.

Secondary

* Explore the association between vitamin D level post-transplant and critical conditions (ICU stay, severity score, infections, mortality).
* Explore the association between vitamin D level post-transplant and pre-transplant conditions (vitamin D level and severity of liver disease).
* Explore the association between pre-transplant vitamin D level and outcome (mortality at 28 days).
* Explore the association between the quality of graft (marginal vs. standard) on post-transplant vitamin D level.
* Explore the association between vitamin D level and graft function.
* Explore the association between post-transplant vitamin D level and long term patient and graft outcomes.

Primary variable end point:

Vitamin D level measured at baseline, and POD (post-operative day) 1, 3, 7, 28. Secondary variable end points ICU length of stay SAPS 2 and SOFA score at POD 1, 7 Days of mechanical ventilation Hospital length of stay Mortality at POD 28 Diagnosed invasive infections Graft rejection in the first 28 days Bilirubin and INR at POD 7 and 28

Data collection and timing of the observations:

Vitamin D level and metabolism:

* Vitamin D at time of listing (wait list for liver transplantation); at time of hospital admission for liver transplantation; POD 1, 3, 7, 28
* Albumin POD 1, 3, 7, 28
* Parathormone (PTH) at time of hospital admission for transplantation, and on 1, 7, 28 SAFETY. Vitamin D levels will be measured in blood samples drawn during standard clinical practice. Clinical activity will follow well established protocols for liver transplants at our institute. Given the observational nature of the study, insurance for possible patient damage is waived.

The patient will be asked for consent to treatment of personal data. The person responsible for this privacy consent will be the principal investigator.

STATISTICAL ANALYSIS. Because this is an exploratory study, all statistical analysis and results will be assessed and reported as exploratory analysis. In order to describe the trend over time of the vitamin D levels in patients undergoing liver transplantation, descriptive statistics such as mean, median, interquartile range and standard deviation will be evaluated. In addition, 95% confidence intervals for mean and standard deviation will be reported. Comparisons between two temporal observations will be assessed with paired t-test.

In addition, mixed model repeated measures (MMRM) will be applied in order to assess the vitamin D trend level over PODs 1-7-28.

In order to assess the secondary aims, the same methods given above will be applied. In particular, for the secondary aim, for the association between quality of graft (marginal vs. standard) on post-transplant vitamin D level, a logistic analysis for repeated measures will be applied.

Any univariate association between factors or covariates, described in the data collection section, will be explored. In addition, multiple MMRM analyses will applied in order to explore association between vitamin D level and the most relevant variables.

All statistical analyses will be done with SAS 9.4, all results will be considered exploratory for statistical testing, and p-values will be reported as "nominally statistically significant." ANALYTICAL METHODS. Vitamin D will be measured with the Bio-Rad 25-OH Vitamin D3/D2 HPLC assay (High Performance Liquid Chromatography). Parathormone will be measured with a chemiluminescence technique using the IMMULITE® 2000 Intact PTH.

ANTICIPATED BENEFITS AND IMPACT OF FINDINGS. Vitamin D deficiency is a global health problem. This study would be an actual description of vitamin D status in a cohort of recipients of liver transplantation, indicating a possible group of patients in which routine measurement of serum vitamin D may be mandatory.

A high prevalence of severe deficiency may suggest starting later high dosage supplementation if new evidence confirms its positive effect in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* All recipients of liver transplantation at Ismett, aged 18 or more

Exclusion Criteria:

* Lack of informed consent for the treatment of personal data. otherwise all the patients will be included if the accept to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study presented in this protocol is the first to focus on vitamin D status in patients undergoing liver transplantation. The primary objective is to study, explore, and describe the level and the trends of vitamin D values over time in liver transplantation recipients in the first days after transplantation, i.e., POD 1, POD 7, and POD 28.
  Because of the lack of knowledge on the association between vitamin D levels and outcomes in this specific cohort no formal sample was calculated beforehand.
  The sample size will be defined by one-year clinical activity: about 60 consecutive patients undergoing liver transplantation will be enrolled during this period.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Describe and explore the level and the trend of vitamin D levels in liver transplantation recipients during the first 28 days after transplantation. | Preoperative and on the post-operative day 28
  Change of the Vitamin D level during the first 28 days after liver transplantation

SECONDARY OUTCOMES:
Explore the association between vitamin D level and critical condition; | Post-operative day 28
  ICU length of stay
Explore the association between pre-transplant vitamin D level and outcome | Post-operative day 28
  Mortality at Post-Operative Day 28
Explore the association between vitamin D level and graft function | Post-operative day 28
  Graft rejection in the first 28 days
Explore the association between vitamin d level and incidence of early post-operative infections | Post.operative day 28
  Diagnosed invasive infections

CONTACTS AND LOCATIONS:
Overall Officials: Gennaro Martucci, MD, Principal Investigator — The Mediterranean Institute for Transplantation and Advanced Specialized Therapies
Locations (1):
- Ismett, Palermo, Italy